CLINICAL TRIAL: NCT01501149
Title: A Randomized Controlled Multi-center Clinical Trial on Treatment of Stage Ⅲ/Ⅳ NK/T Cell Lymphoma With DDGP Regiment (Gemcitabine,Pegaspargase,Cisplatin,Dexamethasone)
Brief Title: Treatment of Natural Killer/T Cell Lymphoma-Ⅲ/Ⅳ
Acronym: CTTNKTL-Ⅲ/Ⅳ
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Collaborators: Second Hospital of Shanxi Medical University (Other); Shanxi Province Cancer Hospital (Other); Wuhan University (Other); Wuhan TongJi Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Qingdao University (Other); Cancer Hospital of Guizhou Province (Other); Xinyang Central Hospital (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2011-2
Record Dates: First submitted 2011-11-29; First posted 2011-12-29 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Nasal and Nasal-type NK/T-cell Lymphoma
Keywords: NK/T cell lymphoma; chemotherapy; clinical trial; RR; PFS; OS
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DDGP regiment (Experimental): DDGP(gemcitabine,pegaspargase,cisplatin,dexamethasone) regiment
  Interventions: Drug: DDGP(cisplatin,dexamethasone,gemcitabine,pegaspargase)
- SMILE Regiment (Experimental): Modified SMILE （methotrexate，hexadecadrol，Ifosfamide，L-AsparaginaseL，Etoposide，Mesna）Regiment
  Interventions: Drug: Modified SMILE （MTX，DEX，IFO，L-ASP，Etoposide，Mesna）

INTERVENTIONS:
Drug: DDGP(cisplatin,dexamethasone,gemcitabine,pegaspargase) — DDP 20 mg/m2,ivgtt（intravenously guttae）,d1-4;DEX 15mg/m2,ivgtt,d1-5;GEM 800mg/m2,ivgtt,30min,d1,8;Pegasparaginase,im,2500IU/m2 d1.Every 21 days for one cycle and three cycles are required. Efficacy was evaluated every two cycles.
  Other Names: DDGP regiment
  Arms: DDGP regiment
Drug: Modified SMILE （MTX，DEX，IFO，L-ASP，Etoposide，Mesna） — MTX,2g/m2 (20% ivgtt（intravenously guttae）,2h;80% ivgtt,4h), d1;DEX,40mg,ivgtt,d2-4;IFO,1.5g/m2,ivgtt,d2-4;L-ASP,6000U/m2,ivgtt,d3-9;VP-16,100mg/m2,ivgtt,d2-4; Mesna,0、4、8h after IFO, 240mg/m2,iv,d2-4.Every 21 days for one cycle and three cycles are required. Efficacy was evaluated every two cycles.
  Other Names: Modified SMILE regiment
  Arms: SMILE Regiment

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of DDGP regiment (gemcitabine，pegaspargase,cisplatin,dexamethasone) for patients with stage Ⅲ/Ⅳ Natural Killer (NK)/T Cell Lymphoma.

DETAILED DESCRIPTION:
Patients with NK/T cell lymphoma usually have a bad prognosis. These patients cannot be treated successfully with the conventional chemotherapy of CHOP. The investigators have been proceeding this trial to evaluate the efficacy and safety of the combination chemotherapy regiment DDGP (gemcitabine，pegaspargase, cisplatin, dexamethasone) in the patients with stage Ⅲ/Ⅳ NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age range 14-70 years old; ECOG performance status 0-2; Estimated survival time > 3 months
* Histological confirmed NK/T cell lymphoma
* None of chemotherapy or radiotherapy has been previously used
* None of chemotherapy contraindication: hemoglobin ≥ 90 g/dl, neutrophil ≥ 1.5×109/L, platelet ≥ 100×109/L, ALT and AST ≤ 2×ULN, serum bilirubin ≤ 1.5×ULN, serum creatine ≤ 1.5×upper limitation of normal (ULN), Serum Albumin ≥ 30g/L, serum plasminogen is normal (Inclusion Criteria of 1,3,6 groups )
* At least one measurable lesion
* None of other serious diseases, cardiopulmonary function is normal
* Pregnancy test of women at reproductive age must be negative
* Patients could be followed up
* None of other relative treatments including the traditional Chinese medicine, immunotherapy,biotherapy except anti-bone metastasis therapy and other symptomatic treatments.
* volunteers who signed informed consent.

Exclusion Criteria:

* Disagreement on blood sample collection
* Patients allergic of any of drug in this regimen or with metabolic disorder
* Pregnant or lactating women
* Serious medical illness likely to interfere with participation
* Serious infection
* Primitive or secondary tumors of central nervous system
* Chemotherapy or radiotherapy contraindication
* The evidence of CNS metastasis
* History of peripheral nervous disorder or dysphrenia
* patients participating in other clinical trials
* patients taking other antitumor drugs
* patients estimated to be unsuitable by investigator

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to end of follow-up-phase (approximately 24 months)

SECONDARY OUTCOMES:
response rate | every 6 weeks,up to completion of treatment(approximately 18 weeks )
  21 days(3 weeks) for one cycle,Efficacy was evaluated every two cycles.
overall survival | up to the date of death (approximately 5 years)
median survival time | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Zhang, Pro，Dr, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Wang X, Zhang L, Liu X, Li X, Li L, Fu X, Sun Z, Wu J, Zhang X, Yan J, Chang Y, Nan F, Zhou Z, Wu X, Tian L, Ma M, Li Z, Yu H, Zhu L, Wang Y, Shi C, Feng X, Li J, Ding M, Zhang J, Dong M, Xue H, Wang J, Zou L, Su L, Wu J, Liu L, Bao H, Zhang L, Guo Y, Guo S, Lu Y, Young KH, Li W, Zhang M. Efficacy and Safety of a Pegasparaginase-Based Chemotherapy Regimen vs an L-asparaginase-Based Chemotherapy Regimen for Newly Diagnosed Advanced Extranodal Natural Killer/T-Cell Lymphoma: A Randomized Clinical Trial. JAMA Oncol. 2022 Jul 1;8(7):1035-1041. doi: 10.1001/jamaoncol.2022.1968. PMID 35708709
- [Derived] Zhao Q, Fan S, Chang Y, Liu X, Li W, Ma Q, Li Y, Wang Y, Zhang L, Zhang M. Clinical efficacy of cisplatin, dexamethasone, gemcitabine and pegaspargase (DDGP) in the initial treatment of advanced stage (stage III-IV) extranodal NK/T-cell lymphoma, and its correlation with Epstein-Barr virus. Cancer Manag Res. 2019 Apr 24;11:3555-3564. doi: 10.2147/CMAR.S191929. eCollection 2019. PMID 31118779
- [Derived] Zhang L, Jia S, Ma Y, Li L, Li X, Wang X, Fu X, Ma W, Qin Y, Li W, Wu J, Sun Z, Zhang X, Nan F, Chang Y, Li Z, Zhang D, Wang G, Yan J, Su L, Wang J, Xue H, Young KH, Zhang M. Efficacy and safety of cisplatin, dexamethasone, gemcitabine and pegaspargase (DDGP) regimen in newly diagnosed, advanced-stage extranodal natural killer/T-cell lymphoma: interim analysis of a phase 4 study NCT01501149. Oncotarget. 2016 Aug 23;7(34):55721-55731. doi: 10.18632/oncotarget.10124. PMID 27384676
- [Derived] Li X, Cui Y, Sun Z, Zhang L, Li L, Wang X, Wu J, Fu X, Ma W, Zhang X, Chang Y, Nan F, Li W, Su L, Wang J, Xue H, Zhang M. DDGP versus SMILE in Newly Diagnosed Advanced Natural Killer/T-Cell Lymphoma: A Randomized Controlled, Multicenter, Open-label Study in China. Clin Cancer Res. 2016 Nov 1;22(21):5223-5228. doi: 10.1158/1078-0432.CCR-16-0153. Epub 2016 Apr 8. PMID 27060152